CLINICAL TRIAL: NCT01057329
Title: Therapeutic Drug Monitoring (TDM) in Child & Adolescent Psychiatry
Brief Title: Therapeutic Drug Monitoring in Child and Adolescent Psychiatry
Acronym: TDMKJP
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Karwautz, Univ. Prof. Dr., Medical University of Vienna
Other Study IDs: 223/2008/TDM; MUW223/2008/2010TDM (Other: MUW); MUW223/2008/2010/TDM (Other: Medical University of Vienna)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Depression; Anorexia Nervosa; ADHD
Keywords: TDM; Drug; Psychopharmacology; children; adolescents
MeSH Terms: conditions — Depression; Anorexia Nervosa; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Duloxetine Hydrochloride; Olanzapine; Aripiprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Anorexia nervosa: 36 severe AN patients treated with aripiprazole
  Interventions: Drug: Aripiprazole
- Anorexia: 36 severe anorexia nervosa patients treated with olanzapine
  Interventions: Drug: Olanzapine; Drug: Aripiprazole
- Attention Deficit Hyperactivity Disorder: 30 ADHD patients treated with atomoxetine
  Interventions: Drug: Atomoxetine
- Depressive disorder: 30 depressed patients treated with duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Atomoxetine — mg according to body weight
  Groups: Attention Deficit Hyperactivity Disorder
Drug: Duloxetine — 30 mg / die
  Groups: Depressive disorder
Drug: Olanzapine — 5mg 1 wwek and 10 mg from second week
  Groups: Anorexia
Drug: Aripiprazole — 5 mg from week 1, 10 mg from week 2
  Groups: Anorexia; Anorexia nervosa

SUMMARY:
The investigators aim to analyse in adolescents with mental illness effectiveness, side effects, and serum level concentrations of antipsychotics (olanzapine and aripiprazole), antidepressants (Duloxetine, Atomoxetine) by means of "Therapeutic Drug Monitoring" (TDM) in order to optimize dosage - effect relations and minimize unwanted side effects.

DETAILED DESCRIPTION:
We aim to analyse in adolescents with mental illness effectiveness, side effects, and serum level concentrations of antipsychotics (olanzapine and aripiprazole), antidepressants (Duloxetine, Atomoxetine) by means of "Therapeutic Drug Monitoring" (TDM) in order to optimize dosage - effect relations and minimize unwanted side effects.

Therapeutic drug monitoring is becoming a quality measure in psychopharmacotherapy in adults and children and has been used successfully recently (Hiemke 2008). In 2007, the German Child & Adolescent Psychiatry University Clinics have founded a network the "TDM-network" headed by Profs. C. Mehler-Wex and J. Fegert in Ulm (www.tdm-kjp-de). The Viennese Child and Adolescent Clinic is part of this network. Most importantly, this network must and wants to be independent from the pharmaceutical industry in order to get un-biased scientific results and data. Within this network, which has been successfully established in the participating clinical departments it is possible to take the lead in several scientific areas.

Highest ethical standards, data-protection and rigorous designs are needed to protect childrens' and adolescents' rights.

Therapeutic drug monitoring (TDM) and its implication for treatment and research: By definition, TDM signifies the dosage of a drug by controlling its concentration in serum. It aims at establishing the therapeutical range of the drug given and thus at minimizing the risk of over- or undermedication (Pschyrembel 2002). Indications for therapeutic drug monitoring in general comprise the following aspects: - Poor response to the administered drug despite a clinically established dosage - Severe side effects despite a clinically established dosage - Combining medications which bear potential to interact adversely with each other - Treatment of patients at risk (immunosuppression, patients in intensive care, patients at need of longterm treatment, patients with a high level of comorbidity or genetic abberations, patients at risk of non-compliance)- Questionable adherence to the treatment regime -Child and adolescent populations

The scientific background of TDM refers to the assumption that the serum concentration of substances along with their active metabolites represent a better measure of their concentration in the brain as the actual dose (Laux & Riederer, 1992; Baumann et al., 2004). Additionally, it is stated that there is a defined relation between serum concentration and clinical effect. This correlation could be confirmed e.g. for the tricyclic antidepressants imipramine und desipramine (Baumann et al., 2004).

Child and Adolescent TDM The psychopharmacotherapy for children and adolescents differs essentially from adults. It is, in its nature, a developmental pharmacotherapy (Herpertz-Dahlmann et al., 2003; Gerlach & Warnke 2004). On a somatic basis, the different developmental stages of children and adolescents, along with their pharmacokinetic variances, don't allow to use similar dosages as in adult patients.

Pharmacokinetics are essentially influenced by body weight, neurophysiological aspects of brain development, a factor which is particularly prone to vulnerability in childhood and adolescence, the gastric milieu and its influence on the uptake of a medication, the frequency of gastric emptying, the development of connective tissue, the proportional distribution of body fat, hormone states, liver metabolism, regulation, expression and function of metabolizing enzymes as well as serum flow in each of the target organs.

Most of the administered drugs, for example, in child and adolescent psychiatry (like tricyclic antidepressants, SSRIs, typical and atypical antipsychotics) are partly or entirely catalyzed via the CYP enzymes, which are localized in the liver. Although genetic expression is limited to the first year of life, regulation and function is largely dependent on the size of organs and their relation to each other as well as to hormone serum concentrations. Thus, these factors are liable to change until the end of puberty.

All these aspects are prone to a much greater variance of side effects and of effects in childhood and adolescence compared to later stages in life (Gerlach et al., 2004).

The vast majority of psychopharmacological agents in child and adolescent psychiatry in Germany is officially not authorized for this age group (Gerlach et al., 2004). Exceptions include, for instance, methylphenidate for the treatment of ADHD or the SSRI fluvoxamine, which can be used for children starting from the age of eight years, for the treatment of obsessive-compulsive disorder.

Since children and adolescents can't be deprived of pharmacotherapy (given the potential major benefits seen in clinical practice and with all experience and data from young adults), the administration of off-label or unlicensed drugs is a practice which is implemented on wide base. As an obvious consequence, safety and efficacy criteria which are established under the Medicines Act, don't apply for the patients of concern. Thus, considerable insecurities among both, medical staff as well as parents (Gerlach & Warnke, 2004), adhere to psychopharmacotherapy in child and adolescent psychiatry.

Addressing the issue of a need for more efficacy and safety in psychopharmacotherapy for youth, TDM in childhood and adolescence does not only provide a general indication for the administration of psychotropic drugs, a field which is largely understudied; it also opens up the opportunity for assessment and clinical response to individually adjust the dosage of drug concentration. Overall TDM intends to make the psychopharmacotherapy more evidence-based and more safe. This is an important issue in this scientific field of medicine which is desideratum long awaited.

From a scientific viewpoint, standardized studies are needed to assess therapeutic ranges of plasma concentrations for children and adolescents. Such studies will give an important insight into the way drugs are metabolized and distributed somatically.

In addition to this, TDM can be considered as a scientifically valid and reliable tool which contributes essentially to the clinical observation of symptom counts and opens up a whole new dimension of data based diagnostics and consequently therapy directives. In this respect, it can be taken as an essential method to improve quality in mental health care among children and adolescents.

We wanted to ensure and enhance qulaity of psychopharmacological treatment in severe anorexia nervosa, ADHD and depression.

ELIGIBILITY:
Inclusion Criteria:

* appropriate diagnosis and severity of the disorder of interest
* age range 10-19

Exclusion Criteria:

* below 10 yrs of age
* no written informed consent possible due to intelligence or no willingness by parents to include minor

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: university clinic population
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Blood level concentrations of the drugs in use; | 5 weeks
  Blood level concentration of the druns in use

SECONDARY OUTCOMES:
Level of symtomatology | 5 weeks
  symtomatology

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karwautz, Prof, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- See also: Eating Disorders and Research Site with links to all projects — http://www.ess-stoerung.eu
- See also: TDM in C&A Psych — http://www.tdm-kjp.de